CLINICAL TRIAL: NCT01774422
Title: Use of the Medical Device DECAP CO2 for the Treatment of Hypercapnic Respiratory Distress in Patients Under Noninvasive Ventilation
Acronym: DECAP CO2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0136; 2012-A01159-34
Record Dates: First submitted 2013-01-07; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Respiratory Distress Syndrome; Hypercapnia
Keywords: Hypercapnia; Respiratory Distress Syndrome; Extracorporeal CO2 remover; Noninvasive ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypercapnia

ARMS (2):
- noninvasive ventilation alone (Experimental): After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:
  * Noninvasive ventilation alone
  * Noninvasive ventilation associated with the DECAP CO2 device
  Interventions: Device: Extracorporeal CO2 removal device
- noninvasive ventilation associated with the DECAP CO2 device (Other): After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:
  * Noninvasive ventilation alone
  * Noninvasive ventilation associated with the DECAP CO2 device
  Interventions: Device: Extracorporeal CO2 removal device

INTERVENTIONS:
Device: Extracorporeal CO2 removal device

SUMMARY:
The patients affected by severe chronic respiratory failure can develop hypercapnic decompensation leading to coma and death in a few hours. At present, the main treatment is noninvasive or invasive ventilation. The noninvasive invasive ventilation requires a minimum of consciousness to insure spontaneous ventilation. In case of noninvasive ventilation impossibility, invasive mechanical ventilation is proposed to patients, which is an aggressive therapy. Regularly, the patients undergo this aggressive therapy without having expressed their opinion. Indeed, a great majority of these patients with severe respiratory insufficiency did not anticipate directives in case of respiratory decompensation (acceptation of aggressive treatments). Efficiency of these aggressive therapies is still uncertain but certainly alters quality of life (discomfort, loss of autonomy…). After complete, clear, loyal and adapted information, a majority of patient do not wish to go on these aggressive therapies. At the time of the decompensation, the patients are incapable to express an opinion because of the hypercapnic narcosis. An extracorporeal CO2 remover device, such as the DECAP CO2, would quickly decrease the hypercapnia what would allow the patient to improve his state of consciousness and so to find the conditions of spontaneous ventilation required for the noninvasive ventilation. The DECAP CO2 device can be used to stop quickly the hypercapnic narcosis and to collect the wills of the patient on the choice of possible aggressive therapies. It is in this last condition that we wish to estimate the DECAP CO2 device.

DETAILED DESCRIPTION:
After validation of the inclusion and exclusion criteria, the patients include in this clinical trial will be randomized between the two arms of the study:

* Noninvasive ventilation alone
* Noninvasive ventilation associated with the DECAP CO2 device

ELIGIBILITY:
Inclusion Criteria:

Adult patient suffering from severe chronic respiratory failure

* Chronic obstructive pulmonary disease : stage III
* Hypercapnic respiratory decomposition
* No anticipated directive with the treating physician, pulmonologist or his family.
* Challenged for invasive ventilation by critical care doctor, emergency doctor or pulmonologist ; due to the respiratory pathology severity or other (age, comorbidity)
* Not challenged for a noninvasive ventilation
* Failure of the noninvasive ventilation in intensive care unit (pH decrease due to hypercapnia after 2 hours of noninvasive ventilation

Obtaining of the consent of the patient or the reliable person or the close relation

Exclusion Criteria:

* - Patients who made anticipated directives (decision of the patient to have no tracheotomy, intubation, noninvasive ventilation)
* Contraindication to heparin (active bleeding, Heparin-induced thrombocytopenia)
* Patients < 18 years and > 90 years
* Patients already included in another therapeutic trial
* Pregnant woman or breast feeding
* Legal incapacity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Hypercapnia | H24

SECONDARY OUTCOMES:
Blood gases | H0
Duration of judgment disability | H72
Duration of blood pH normalization | H72
Duration of hypercapnia | H72
Glasgow | H0
SAPSII scores(Simplified Acute Physiology Score II) | H24
Duration of noninvasive ventilation | H72
Duration of hospitalization | H72
Mortality | H72
MMSE (Mini Mental State Examination) | H0
ACE ( Aid To Capacity Evaluation)scores | H0
SOFA scores(Sepsis-related Organ ) | H24
Blood gases | H1
Blood gases | H2
Blood gases | H3
Blood gases | H4
Blood gases | H6
Blood gases | H12
Blood gases | H18
Blood Gases | H24
Blood gases | H32
Blood gases | H40
Blood gases | H48
Blood gases | H56
Blood gases | H64
Blood gases | H72
Glasgow | H4
Glasgow | H8
Glasgow | H24
Glasgow | H36
Glasgow | H48
MMSE (Mini Mental State Examination) | H4
MMSE (Mini Mental State Examination) | H8
MMSE (Mini Mental State Examination) | H24
MMSE (Mini Mental State Examination) | H36
MMSE (Mini Mental State Examination) | H48
ACE ( Aid To Capacity Evaluation)scores | H4
ACE ( Aid To Capacity Evaluation)scores | H8
ACE ( Aid To Capacity Evaluation)scores | H24
ACE ( Aid To Capacity Evaluation)scores | H36
ACE ( Aid To Capacity Evaluation)scores | H48

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAUTRETTE, Principal Investigator — University Hospital, Clermont-Ferrand